CLINICAL TRIAL: NCT04019470
Title: Immunomodulation Analysis on Peripheral Blood Mononuclear Cells of Radiation Therapy in Pediatric Malignant Brain Tumors
Brief Title: Immunomodulation Analysis of Radiation Therapy in Pediatric Malignant Brain Tumors
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Cancer Center Director, Capital Medical University
Other Study IDs: IRPBT
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Brain Tumor, Pediatric
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the effect of radiotherapy on peripheral blood immune cell composition and function in pediatric malignant brain tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* Age from 3 to 18
* To be diagnosed with malignant brain tumors
* To eligible for radiation therapy
* Karnofsky performance status ≥ 70
* No prior radiation exposure
* Informed consent signed for blood sample collection and used for research purpose

Exclusion Criteria:

* Patients had received radiotherapy previously.
* Patients who had no histological diagnosis
* Patients who do not wish to participate
* Patients with infections

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The brain tumors patients between the ages of 3 year and 18 years who will be received radiation therapy evaluated and determined by their physician
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
The changes of peripheral blood immune cells | 6 weeks (prior and post the radiation therapy )
  The flow cytometric analysis of lymphocyte subtypes populations would be performed

SECONDARY OUTCOMES:
Activation status of T cells | 6 weeks (prior and post the radiation therapy )
  Activation status of peripheral IFN-γ-producing effector CD8+ T cells by Elispot.
The changs of inflammatory cytokines and chemokines | 6 weeks (prior and post the radiation therapy )
  Human inflammatory cytokines and chemokines will be analyzed by ELISA during radiation therapy. The cytokines and chemokines are IL-2, IL-10, IFN-γ, TNF-α

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital Cancer Center, Beijing, China